CLINICAL TRIAL: NCT00300209
Title: Manhattan HIV/Hepatology Brain Bank
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 98-0477; R24MH059724 (NIH)
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: HIV; Hepatitis
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum blood

SUMMARY:
Description: The Manhattan HIV/Hepatology Brain Bank (MHBB) was established in 1998 as a resource for the AIDS research community. The MHBB was created to act as a center for the provision of pre- and post-mortem tissues and body fluids from HIV infected persons. It has recently expanded its goals to assist in the elucidation of liver disease-induced nervous system disorders.

The MHBB is dedicated to improving the understanding of HIV and Hepatitis C and thereby, improving the lives of patients living with HIV and/or Hepatitis C.

Participation is voluntary and can be stopped at any time.

Benefits: This is an observational study; no experimental procedures, devices or drugs are used. All enrolled patients undergo regular examinations by physicians, nurses, and neuropsychologists who specialize in the problems that HIV and HCV can cause.

Taking part in this study may result in the detection of brain, muscle, or spinal cord disease for which treatments may be available. Participants may receive no direct benefit from this study. However, knowledge gained from this research may, in the future, help others who suffer from HIV/AIDS and/or liver disease.

Participants agree to autopsy and organ donation upon demise by signing an Anatomical Gift Consent document.

ELIGIBILITY:
Inclusion Criteria:

CD4 < 50 on two occasions >12 weeks apart. Hemoglobin <10 G/dL. Albumin <3.2 G/dL.

CMV end-organ disease Disseminated MAC PML AIDS Dementia Complex Wasting (>30% of lean body mass)

Visceral Kaposi's sarcoma Lymphoma-systemic of CNS

CHF Major systemic illness with poor prognosis (as determined by primary physician).

Exclusion Criteria:

- <18 years old Not willing to sign an Anatomical Gift Consent for autopsy and organ donation upon demise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HIV infection with advanced disease who display signs of distal sensory polyneuropathy, and who consent to postmortem organ donation.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 1998-09; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Viral Load blood level | Baseline
  Plasma viral load level

SECONDARY OUTCOMES:
CD4 cell blood level | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Susan Morgello, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Result] Morgello S, Estanislao L, Simpson D, Geraci A, DiRocco A, Gerits P, Ryan E, Yakoushina T, Khan S, Mahboob R, Naseer M, Dorfman D, Sharp V; Manhattan HIV Brain Bank. HIV-associated distal sensory polyneuropathy in the era of highly active antiretroviral therapy: the Manhattan HIV Brain Bank. Arch Neurol. 2004 Apr;61(4):546-51. doi: 10.1001/archneur.61.4.546. PMID 15096404